CLINICAL TRIAL: NCT03755648
Title: Effect of Delorme Resistance Exercises Versus Treadmill Training on Locomotor Abilities in Cerebral Palsy
Brief Title: Effect of Delorme Resistance Exercises Versus Treadmill Training in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Principal Investigator, Samreen Sadiq, Principal Investigator, Ghurki Trust and Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2018-11-09; First posted 2018-11-28 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
Keywords: Delorme resistance exercises; treadmill training; locomotor abilities; tendon of achilles lengthening
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treadmill training (Experimental): Group A: received treadmill training along with traditional physiotherapy.. The motorized treadmill was used keeping treatment parameters as 50 Hertz, 10 Ampere and 220 Volts The treadmill training was provided by giving instructions first and then warm up was given for 5 minutes prior to the training. The children were upright with the feet flat on treadmill platform. The height of handrails was adjustable according to every child thus keeping their gaze forward. The training was ended at cool down period of 5 minutes
  Interventions: Other: Treadmill training
- traditional physical therapy (Other): Traditional therapy includes use of hot packs for 15 minutes and stretching for 20 minutes which will be applied to both groups prior to actual intervention
  Interventions: Other: traditional physical therapy
- Delorme Resistance exercise (Experimental): Group B received delorme resistance exercise with traditional physiotherapy. Delorme Resistance Training was also initiated with 5 minute warm up period. It was started with 10 Repetition Maximum and was gradually increased. The treatment session was thirty minutes for each group, six times a week for three months.
  Interventions: Other: Delorme resistance exercise

INTERVENTIONS:
Other: Treadmill training — The motorized treadmill treatment parameters considered will be 50 Hertz, 10 Ampere and 220 Volts. The speed of treadmill will be controlled with a single finger tip allowing an individual to exercise in safe environment with sufficient space.The treadmill training will be provided by giving instructions first and then warm up will be given for 5 minutes prior to the training. The children will be upright with the feet flat on treadmill platform. The height of handrails will be adjustable according to every child thus keeping their gaze forward. The training will be ended at cool down period of 5 minutes.The treatment session will be thirty minutes for each group, six times a week for three months.
  Other Names: traditional physical therapy
  Arms: Treadmill training
Other: traditional physical therapy — Traditional therapy includes hot pack for 15 minutes and stretching for 20 minutes
  Arms: traditional physical therapy
Other: Delorme resistance exercise — Delorme Resistance Training was also initiated with 5 minute warm up period. It was started with 10 Repetition Maximum and was gradually increased. The treatment session was thirty minutes for each group, six times a week for three months.
  Other Names: traditional physical therapy
  Arms: Delorme Resistance exercise

SUMMARY:
Cerebral palsy is one of the most important source of disability among children and its incidence is almost 3.6 in thousand live births.Children with Cerebral Palsy presents with ambulatory difficulties.The current study highlights the effect of treadmill training as compared to DeLorme resistance exercises on locomotor activities in cerebral palsy child.The present study would add to the clinical knowledge of physical therapists by promoting the implementation of treadmill training and DeLorme resistance exercises for this prevalent pediatric neurodevelopmental disorder. The study would decrease the burden of disease among community and enhance the social participation of cerebral palsy children. This in turn would improve the quality of living of these disabling diseased children.

ELIGIBILITY:
Inclusion Criteria:

* Children with Gross Motor Functional Scale Level II and III
* Ability to understand commands and directions
* Diplegic type of cerebral palsy
* Children who had undergone bilateral Tendon of Achilles Lengthening procedure 3 to 6 months post-operatively

Exclusion Criteria:

* Children presenting with other types of Cerebral Palsy
* Children with audiovisual impairment that can hinder the treatment
* leg length discrepancy greater than 2 cm,
* Fixed contractures, joint instability and associated cardiovascular condition.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Locomotor ability | 1 month
  Locomotor ability was assessed using ABILOCO-kids questionnaire. It consisted of 10 locomotion activities of which difficulty was rated by the parents. It has good reliability r=0.97 and reproducibility of 0.96. Parent is asked to fill in questionnaire by estimating their child's ease or difficulty in performing each activity. Activities are presented in 10 different random orders to avoid any systematic effect. During evaluation, 3-level response scale is presented to parent. Parent is asked to rate his perception on response scale as 'Impossible', 'Difficult' or 'Easy'. Activities not attempted by child within last 3 months are not scored and are entered as not applicable. Activities that child doesn't perform because they are too difficult must be scored as 'Impossible'. Child's locomotion ability and its 95% confidence interval are located on locomotion ability scale expressed in logits. Higher the ability of a child the more the measure will be located to the right.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz Asim, DPT (USA), Study Chair — Lahore Medical and Dental college
Locations (1):
- Samreen Sadiq, Lahore, Punjab Province, Pakistan

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03755648/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03755648/SAP_003.pdf